CLINICAL TRIAL: NCT02189655
Title: Diluting With Cerebrospinal Fluid Versus Traditional Intrathecal Administration: Antishivering Effects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Department of Anesthesiology, The First Hospital of CMU, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20140630
Record Dates: First submitted 2014-06-30; First posted 2014-07-14 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Antishivering Effects
Keywords: shivering spinal anesthesia
MeSH Terms: interventions — Bupivacaine; Indicator Dilution Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Control (No Intervention): Hyperbaric bupivacaine 0.5% 2.5 mL was administered intrathecally in 30 seconds.
- Group Diluting with cerebrospinal fluid (Experimental): Hyperbaric bupivacaine 0.5% 2.5 mL diluting with cerebrospinal fluid was administered intrathecally in 30 seconds
  Interventions: Procedure: bupivacaine 0.5% 2.5 mL diluting with cerebrospinal fluid

INTERVENTIONS:
Procedure: bupivacaine 0.5% 2.5 mL diluting with cerebrospinal fluid — Hyperbaric bupivacaine 0.5% 2.5 mL diluting with cerebrospinal fluid was administered intrathecally in 30 seconds
  Arms: Group Diluting with cerebrospinal fluid

SUMMARY:
This prospective randomized double-blinded study was conducted to compare the antishivering effects of two different types of intrathecal administration.

DETAILED DESCRIPTION:
This prospective randomized double-blinded study was conducted to compare the antishivering effects of two different types of intrathecal administration.Group Control:traditional intrathecal administration; Group Diluting:Diluting with cerebrospinal fluid

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status Ⅰ or Ⅱ who were scheduled for elective surgery under spinal anesthesia were enrolled.

Exclusion Criteria:

* Patients with pre-operative fever (>38℃), diabetes, , Parkinson's disease, hypo or hyperthyroidism, Raynaud's syndrome, obese patients (weight >100 kg), patients shorter than 152 cm, those with a history of allergy to the study medications, and patients receiving vasodilators were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
antishivering effects of two different types of spinal anesthesia | time point 1: 15 minuntes after spinal anesthesia and time point 2 : when patiets were sent to postoperation care unit
  antishivering effects of two different types administration of spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ma, M.D.,Ph.D, Study Director — The First Hospital of CMU
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China